CLINICAL TRIAL: NCT06465394
Title: Exercise-induced Hypoalgesia and Proprioceptive Changes, Comparing Isometric to Isotonic Neck Exercises
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Dakota (Other)
Responsible Party: Principal Investigator, Kory Zimney, PT, DPT, PhD, Associate Professor, University of South Dakota
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-24-100
Record Dates: First submitted 2024-06-10; First posted 2024-06-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric Exercise (Active Comparator): Isometric test protocol. Participants will be asked to perform the exercise at a moderate exercise level (3/10 on the mRPE scale provided to them). They will complete a 1, 10-second isometric hold to their hand dominant side (if ambidextrous, the side the participant would report as the most dominant side) to allow them to find their "moderate" intensity level. The participant will then take a 2-minute rest before beginning the exercise routine and will be instructed to keep a consistent resistance level during the exercise bout. During the exercise, the subjects will hold the rotation contraction for 10 seconds, take a 2-second rest, complete this 5 times, and then change to the left side. They will do this for 3 sets of right and left. Researchers will time the exercises and give verbal instructions to make sure they are performing for the appropriate amount of time and rest periods.
  Interventions: Procedure: Exercise
- Isotonic Exercise (Active Comparator): The resistance level will stay at the participant's selected moderate level during the entire testing unless they need to stop due to pain or difficulty completing the exercise. During the exercise, the participants will be rotating to the right first at a pace of 1 second for concentric contraction to full rotation and 1 second for eccentric contraction, returning the head to the neutral position. The participant will continue this pace to complete 5 repetitions and then take a 2-second rest before continuing this sequence 5 times (a total of 25 reps) before switching and doing left rotation in the same fashion. This will be done for a total of 3 sets for both right and left rotation. The use of a metronome will be used along with the researcher's verbal instructions and cueing to maintain the proper sequence and timing of the exercise.
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — Neck exercises in a cross over design that the participants will do both types of interventions with a washout period inbetween.

SUMMARY:
Exercised induced hypoalgesia (EIH) (reduction in pain) after exercise has been studied in the literature, but no comparisons have been made specifically looking at different types of exercise (isometric/dynamic moving through a range of motion with resistance versus isotonic/applying static resistance to a joint not moving) with neck muscle strengthening. This study will explore to see if one form of exercise is superior to the other in providing EIH.

Another benefit of exercise is improving proprioception (knowing where our body is in space). Again no specific investigation has been done comparing isometric versus isotonic exercises for neck muscles.

Both of these exercises are often prescribed in physical therapy so further understanding the benefits of them can help improve the prescription of exercises for patients.

DETAILED DESCRIPTION:
After consent has been obtained, participants will be asked the screening questions to confirm eligibility for the study. The researcher will then ask the participants demographic questions and record the responses for age, gender, racial category, and handedness. Odd-numbered participants will perform isometric exercises first and then isotonic exercises on the second day. Even numbered participants will perform isotonic exercises first and then isometric exercises on the second day. There will be 2-3 days between each test period. Testing each time will have participants do baseline measurements for pain pressure threshold (PPT) and proprioception (JPE), exercise protocol, and then retest PPT and JPE post exercise.

Pain pressure threshold testing consists of measuring the distance between C7 and the distal aspect of the acromion while the participant is seated. If possible, the shirt will be removed for men, or the neck color pulled to the side for females. If unable to move the shirt to the side, the testing can be done over the clothing. The mid-way point will be marked with a pen or other method to indicate the location on the upper trap muscle where the PPT testing will be performed on both the right and left sides. Utilization of a pressure algometer will be used for testing with a 1 cm2 rubber tip. The pressure algometer tip will be placed on the mark of the midpoint of the upper trap previously measured and marked. Pressure is slowly applied until the participant reports a change from pressure to pain and says "STOP". At the moment the participant says stop, the pressure is stopped, and the recording is measured. There will be 3 tests with PPT on both right and left alternating between each side with testing.

Proprioception is measured by the joint position error (JPE) test. This test requires the patient to place a headlamp equipped with a laser pointer. They will be seated in a chair facing a wall with the JPE target on the wall. The subject is to sit with their head in a normal resting state, looking straight ahead. The target is adjusted to the participant's baseline. The participant is instructed to get a "sense" of this position. The participant then moves their head/neck to the right or left, returning to their resting position. The subject then closes their eyes and completed 6 trials of turning their head to the right and 6 trials to the left. The researcher will assist them in recentering to their start position each time before the next rotation of the head/neck.

Once the baseline PPT and JPE are measured, the subjects will go through the exercise protocol.

Isometric test protocol. Participants will be asked to perform the exercise at a moderate exercise level (3/10 on the mRPE scale provided to them). They will complete a 1, 10-second isometric hold to their hand dominant side (if ambidextrous, the side the participant would report as the most dominant side) to allow them to find their "moderate" intensity level. The participant will then take a 2-minute rest before beginning the exercise routine and will be instructed to keep a consistent resistance level during the exercise bout. During the exercise, the subjects will hold the rotation contraction for 10 seconds, take a 2-second rest, complete this 5 times, and then change to the left side. They will do this for 3 sets of right and left. Researchers will time the exercises and give verbal instructions to make sure they are performing for the appropriate amount of time and rest periods. After completing the exercise protocol, they will complete the PPT and JPE tests in the same way as was done for baseline measurement.

Isotonic test protocol. Participants will be asked to perform the exercise at a moderate exercise level (3/10) on the mRPE scale provided to them). They will complete 2 reps using the red rubber band resistance on the 'NecksLevel' neck strengthening device, moving through a full range of motion toward their hand-dominant side as they will do in the isometric test. After completing the 2 test reps, they will be asked if they would like to increase or decrease the resistance to be at a moderate level. The new resistance level or staying the same level will then be done for 3 more reps to ensure they are at a moderate level. The participants will then take a 2-minute rest before beginning the exercise routine. The resistance level will stay at the participant's selected moderate level during the entire testing unless they need to stop due to pain or difficulty completing the exercise. During the exercise, the participants will be rotating to the right first at a pace of 1 second for concentric contraction to full rotation and 1 second for eccentric contraction, returning the head to the neutral position. The participant will continue this pace to complete 5 repetitions and then take a 2-second rest before continuing this sequence 5 times (a total of 25 reps) before switching and doing left rotation in the same fashion. This will be done for a total of 3 sets for both right and left rotation. The use of a metronome will be used along with the researcher's verbal instructions and cueing to maintain the proper sequence and timing of the exercise. After completing the exercise protocol, they will complete the PPT and JPE tests in the same way as was done for baseline measurement.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old,
* all genders,
* healthy individuals with no neck pain

Exclusion Criteria:

* Medical restrictions to physical activity
* History of chronic pain (pain > 3 months) or current acute neck pain
* Unable to refrain from alcohol, pain medications, and vigorous exercise 24 hours prior to testing

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
PPT | Pre post measure before and after exercise session taking approximately 10 minutes
  Pain Pressure Threshold with use of algometer

SECONDARY OUTCOMES:
JPE | Pre post measure before and after exercise session taking approximately 10 minutes
  Joint position error utilizing measurement in cm from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kory J Zimney, PhD, Principal Investigator — University of South Dakota
Locations (1):
- University of South Dakota, Vermillion, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No